CLINICAL TRIAL: NCT00684229
Title: Regional Anesthesia in Patients Undergoing Colon-Rectal Surgery
Brief Title: Regional Anesthesia in Colon Rectal Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: investigator could not identify any patients
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Andrea Kurz, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 07-933
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Colon Cancer
Keywords: Anesthesia; regional; Cancer recurrence; Anesthesia; inhalational; Analgesia; opioid
MeSH Terms: conditions — Colonic Neoplasms; Agnosia | interventions — Anesthesia, Conduction; Analgesia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regional anesthesia and analgesia (Active Comparator): Regional anesthesia and analgesia (either epidural or paravertebral anesthesia).
  Interventions: Procedure: Regional anesthesia and analgesia
- general anesthesia followed by opioid analgesia (Active Comparator): Subjects randomized to arm 2 will receive general anesthesia followed by opioid analgesia.
  Interventions: Drug: general anesthesia followed by opioid analgesia

INTERVENTIONS:
Procedure: Regional anesthesia and analgesia — Post-operative analgesia will be epidural bupivacaine and fentanyl as well as intravenous morphine.
  Arms: Regional anesthesia and analgesia
Drug: general anesthesia followed by opioid analgesia — sevoflurane general anesthesia and postoperative opioid analgesia
  Arms: general anesthesia followed by opioid analgesia

SUMMARY:
This study will compare recurrence rates in patients with colorectal cancer who will be randomly assigned to epidural anesthesia/analgesia combined with general anesthesia or to general anesthesia followed by opioid analgesia.

DETAILED DESCRIPTION:
The study population will consist of patients who are scheduled for open laparoscopic or laparoscopic assisted surgery for colon cancer. Patients will randomized into one of two groups. The intervention group will receive combined regional and general anesthesia during surgery. Postoperative pain treatment will be based on regional anesthesia techniques. The Control group will receive general anesthesia during surgery. Postoperative pain treatment will be based primarily on opioids. After surgery, patients will be followed daily during their hospital stay. Patients will be contacted by telephone every 6 months for five years. Quality of life questionnaires will be administered at these follow ups.

ELIGIBILITY:
Inclusion Criteria:

* Primary colon cancer without known extension beyond colon (T3, N0, M0)
* Scheduled for open, laparoscopic assisted and laparoscopic resection of the colon.
* Written informed consent, including willingness to be randomized to epidural anesthesia/analgesia or to sevoflurane general anesthesia and postoperative opioid analgesia.

Exclusion Criteria:

* Previous surgery for colon cancer;
* Any contraindication to epidural anesthesia or analgesia (including coagulopathy, abnormal anatomy);
* Any contraindication to midazolam, propofol, sevoflurane, fentanyl, or morphine;
* Age <18 or >85 years old;
* ASA Physical Status ≥4;
* Other cancer not believed by the attending surgeon to be in long-term remission;
* Systemic disease believed by the attending surgeon or anesthesiologist to present ≥25% two-year mortality.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
cancer recurrence | 5 years
  To determine if recurrence of local/metastatic cancer after open and laparoscopic resection colon cancers is lower in patients randomized to epidural anesthesia & analgesia than to sevoflurane general anesthesia and postoperative opioid analgesia

SECONDARY OUTCOMES:
length of post operative hospitalization | days
  To determine if the length of post operative hospitalization is shortened in patients randomized to epidural anesthesia & analgesia than to sevoflurane general anesthesia and postoperative opioid analgesia.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Sessler, MD, Study Chair — The Cleveland Clinic; Andrea Kurz, MD, Principal Investigator — The Cleveland Clinic
Locations (3):
- Cleveland Clinic, Cleveland, Ohio, United States
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina
- University of Dusseldorf, Düsseldorf, Germany